CLINICAL TRIAL: NCT00166946
Title: Effects of Arsenic on Keratinocytes in a Skin Equivalent Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 9361701179
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-12-21 (Estimated); Status verified 2004-11

CONDITIONS: Bowen Disease
MeSH Terms: conditions — Bowen's Disease | interventions — Microphysiological Systems

INTERVENTIONS:
Procedure: foreskin from healthy adults for organotypic culture

SUMMARY:
We popose that arsenic-induced lymphocytes dysfunction plays an important role in biological mechanisms of arsenical Bowen's disease.

DETAILED DESCRIPTION:
Arsenical cancers (comprising skin, bladder, kidney, lung, colon and liver malignancies) were prevalent in southwestern coast of Taiwan where the artesian water was contaminated with high concentration of arsenic. Skin is a main target of arsenical poisoning. The cutaneous manifestations of chronic arsenism can take form as hyperpigmentation, hypopigmentation, arsenical keratosis and arsenical skin cancers. The most popular arsenical skin cancer is Bowen's disease, which is a carcinoma in situ of skin and often confined to sun-protected skin. Pathologically, there are several characteristics present in Bowen's disease: (1) abnormal cell proliferation and carcinogenesis in keratinocytes; (2) dysplasia and apoptosis at the lesion; (3) integrin deficiency/defect in the basal cells of the skin; (4) dysfunctions in peripheral immune cells. Our pervious results indicated that arsenic affected cell cycle regulation by influencing the proliferation and apoptosis of keratinocytes. Furthermore, we found that integrins were deficient in basal layer of lesional and perilesional sites of Bowen's disease as demonstrated by immunohistochemistry. The integrin deficiency in Bowen's disease might lead to abnormality of cell cycle regulation, differentiation and carcinogenesis. In addition, arsenic can destruct lymphocytes to cytokine regulation and induce lymphocytes apoptosis. We propose that arsenic-induced lymphocytes dysfunction plays an important role in biological mechanisms of arsenical Bowen's disease. There are many regulatory mechanisms involved in progression of chemical carcinogenesis, including the reactions among carcinogen and target cells, supporting cells and immune interactions. Therefore, this study is to investigate these skin cell-cell interactions induced by arsenic using an organotypic epidermis culture model. By using this model, we can mimic the mechanism of arsenic-induced skin diseases. Which will give us much more information that similar to carcinogenesis progesee in human body as compared to cell culture model. The effects of arsenic on epidermis formation, the effects of UVB and arsenic on arsenical carcinogenesis and the interactions between immune cells and skin cells will be studied in this 3-year proposal as described below:

The 1st year: Study of arsenical effects on integrin expression, cell proliferation, differentiation and apoptosis in organotypic epidermis.

The 2nd year: Study of arsenic and/or UVB -induced biological changes in organotypic epidermis and Bowen's disease.

The 3rd year: Study of the interactions between immune cells and epidermal cells induced by arsenic.

This study will give us much more information that similar to carcinogenesis progesee in human body as compaired to cell culture model. We hope the result of this study can provide a useful model in chemical carcinogenesis investigation field.

ELIGIBILITY:
Inclusion Criteria:

Normal healthy adult -

Exclusion Criteria:

systemic disease or with a history of exposure to arsenic-

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2005-06; Study Completion 2008-01

PRIMARY OUTCOMES:
we collect foreskin from healthy adults

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Su Yu, MD PHD, Study Director — National Taiwan Univesity Hospital, Dept. of Dermatology
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei, Taiwan, Province of China
  - National Taiwan University Hospital, Taipei